Feeling and Body Investigators for Pediatric Abdominal Pain (FBI)

NCT02075437

01/28/2019

## Primary Outcome 1. Percentage of Participants Who Complete Treatment

Participants were considered to have completed treatment if they completed all 10 treatment sessions.

## Primary Outcome 2. Percentage of Participants Completing Homework Assignment

As part of the study, participants were asked to complete homework assignments after each treatment session. These assignments consisted of weekly pain diaries, which included both parent reports of child experience and child reports of their own experience of different types of pain. At pre-treatment and post treatment these parent and child ratings were completed three times daily (beginning of day, before dinner, and end of day), with the end of day assessments asking about the worst pain that day and the others assessing pain at that moment. For homework assignments given during treatment sessions, participants were asked only to report at one time point (end of day) daily.

• In assessing participants' completion rate of their homework assignments all pain diaries were entered into a singular database, and reverified to ensure data quality control. Once all data was collected, all weekly pain diaries were assessed for completion and given a label indicating their level of completion, the labels and criteria are described below.

| Label | Meaning |
|---|---|
| Complete | Participant completed all days of the end of day diary packet |
| Complete Partial | Participant completed 4 or more days of the end of day diary packet |
| Incomplete Partial | Participant completed 3 or less days of the end of day diary packet |
| Not Completed | Participant did not complete any days in the end of day diary packet |
| Not Given | Participant not given end of day diary packet |

- For our analysis, if a participant completed at least 1 pain diary entry in a weekly pain diary they were considered as having successfully completed their homework assignment for that given week.
- Once all participant labeling was completed percentages of completion rates were calculated by dividing the number of homework completions by the number of homework assignments given. Those with a completion percentage of equal or greater than 90% were then considered to be "successful".